CLINICAL TRIAL: NCT05735912
Title: Endoscopic Ultrasound-guided RAdiofrequency Ablation Versus Surgical Resection for the Treatment of Pancreatic INsulinoma: a Multicenter Randomized Controlled Trial
Brief Title: EUS-RFA Versus Surgery for Pancreatic Insulinoma (ERASIN-RCT)
Acronym: ERASIN-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Stefano Francesco Crinò, MD, Doctor, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4121CESC
Record Dates: First submitted 2023-02-01; First posted 2023-02-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Insulinoma
MeSH Terms: conditions — Insulinoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic ultrasound-guided radiofrequency ablation (Experimental): Endoscopic ultrasound-guided radiofrequency ablation will be performed using the "EUSRA" system (Taewoong, Seoul, Korea). The system consists of a 19-gauge needle electrode (140-cm long), a radiofrequency current generator (VIVA RF generator; Taewoong), and an inner cooling system that circulates chilled saline solution during the radiofrequency ablation procedure. The inner metal part is insulated over its entire length, with the exception of the terminal 5 to 20mm for energy delivery. The needle electrode is attached to the radiofrequency current generator and to a cooling pump. The generator, in addition to providing radiofrequency current, allows the control of physical power and impedance parameters.
  Interventions: Procedure: Endoscopic ultrasound-guided radio frequency ablation
- Surgery (Active Comparator): Surgical resection will be performed in an inpatient setting. The type and extension of surgical resection, as well as need for lymphadenectomy, will be decided by the treating surgeons according to the tumor position, distance from the main pancreatic duct, and local expertise.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided radio frequency ablation — Radiofrequency ablation performed under endoscopic ultrasound guidance of pancreatic insulinoma
  Arms: Endoscopic ultrasound-guided radiofrequency ablation
Procedure: Surgery — Surgical resection of pancreatic insulinoma
  Arms: Surgery

SUMMARY:
The goal of this muticentre randomized controlled trial is to compare endoscopic ultrasound-guided radiofrequency ablation (EUS-RFA) with surgery for treatment of pancreatic insulinoma. The main questions it aims to answer are: 1) What is the safest treatment? 2) Is efficacy comparable? Patients will be randomized to undergo EUS-RFA or surgical resection. Researchers will compare the rate of adverse events and the clinical efficacy after the two treatments to see if EUS-RFA result safer and effective compare with surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of pancreatic insulinoma (38) (e.g., fasting test, insulin blood levels, C-peptide blood levels)
* Presence of a visible single pancreatic nodule on imaging (computed tomography, and/or magnetic resonance imaging, and/or endoscopic ultrasound).
* No evidence of distant localizations visualized at computed tomography, and/or magnetic resonance imaging, and/or endoscopic ultrasound
* Tumor ≤ 2cm
* Informed consent provided by the patient or closest relative.

Exclusion Criteria:

* G2 with Ki-67 >5% on histological examination at EUS-guided biopsy samples (if performed)
* Distance between lesion and main pancreatic duct ≤ 1mm or upstream dilation of the main pancreatic duct
* Metastatic tumor at the time of diagnosis
* Multiple pancreatic nodules
* Diagnosis of multiple endocrine neoplasia type 1 according to guidelines
* Unfit for surgery or high-risk surgical patients
* Endoscopic ultrasound not feasible for surgical altered anatomy
* Known bleeding disorder that cannot be sufficiently corrected with co-fact or fresh frozen plasma
* Use of anticoagulants that cannot be discontinued
* International normalized ratio >1.5 or platelet count <50.000
* Pregnancy or breast feeding
* Failure to sign the patient's or closest relative's informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | Up to 72 months
  Rate of overall and severe adverse events will be recorded

SECONDARY OUTCOMES:
Clinical effectiveness | Up to 72 months
  Rate of patients experiencing symptoms disappearance
Evaluation of quality of life by questionnaire | Up to 72 months
  Assessment of quality of life using a questionnaire
Length of hospital stay | Up to 72 months
  Days of hospitalization
Recurrence | Up to 72 months
  Rate of local or distant recurrence
Reintervention | Up to 72 months
  Rate of reintervention
Pancreatic insufficiency | Up to 72 months
  Rate of endocrine or exocrine pancreatic insufficiency

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Verona, Verona, Italy